CLINICAL TRIAL: NCT05343221
Title: The Effect of Haptic and Highly Fidelity Simulator Use on Knowledge, Skills, Satisfaction and Self-Confidence Levels in Cardiopulmonary Resuscitation Training: A Randomized Controlled Study
Brief Title: The Effect of Haptic and Highly Fidelity Simulator in Cardiopulmonary Resuscitation Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, İlayda Türkoğlu, Lecturer at the Nursing Faculty and co-researcher, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E-46418926-050.01.04--84464
Record Dates: First submitted 2022-04-09; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Nursing Caries; Cardiopulmonary Resuscitation
Keywords: Haptic; Highly Fidelity Simulator; Skills; Satisfaction; Training
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: This study will conducted between April and July 2022 on 60 volunteer students studying in the Department of Nursing Faculty in Turkey. The inclusion criteria were as follows being 18 years old or over, being a fourth year student, be in the classroom on training day. The students included in the study were randomly divided into two groups.The Haptic group will use the Haptic Device with 3D technology and the High Fidelity Simulator group will use High Fidelity CPR Simulator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haptic (Experimental): Practice in Haptic Group: Students will be taught cardiopulmonary resuscitation skills with the 3D Systems Touch Haptic Simulator. During the application, there will be 2 researchers and the student who made the application in the room. While one of the researchers will be with the student only for support during the practice, the other researcher will fill the "Cardiopulmonary Resuscitation Skills Checklist" by evaluating the cardiopulmonary resuscitation skill of the student.
  Interventions: Device: Haptic
- High Fidelity Simulator (Experimental): Application in the Simulator Group with High Fidelity: Students will be taught cardiopulmonary resuscitation skills with the CPR Simulator. The student and 2 researchers who will practice will remain in the environment, and the student will also be asked to practice.
  Interventions: Device: High Fidelity Simulator

INTERVENTIONS:
Device: High Fidelity Simulator — First of all, students will be given 1 hour of CPR training. Then they will be asked to apply with the High Fidelity CPR Simulator. This simulator is adult human sized and specialized for CPR practice. It will not be interfered during the application. The student's practice will be evaluated by an observer. The student will evaluate his/her satisfaction after the application is over.
  Arms: High Fidelity Simulator
Device: Haptic — First of all, students will be given 1 hour of CPR training. Then they will be asked to apply with the 3D technology Haptic Device Simulator. This tool has a computer screen and a swing haptic pen. It will not be interfered during the application. The student's practice will be evaluated by an observer. The student will evaluate his/her satisfaction after the application is over.
  Arms: Haptic

SUMMARY:
Cardiopulmonary Resuscitation (CPR) is of great importance for nurses who frequently encounter cardiopulmonary arrest in health care institutions and who are within their duties, authorities and responsibilities. Therefore, nurses should have sufficient, up-to-date knowledge and skills about cardiopulmonary resuscitation. Nursing educators should try different training methods on CPR education and ensure that the student has sufficient knowledge and skills before graduation. This study, In order to examine the effects of haptic and highly fidelity simulator use in Cardiopulmonary Resuscitation training in nursing students on their knowledge, skills, satisfaction and self-confidence levels, it was planned to be performed in a randomized controlled type.

DETAILED DESCRIPTION:
This study aim to examine the effects of Haptic and Highly Fidelity Simulator use in Cardiopulmonary Resuscitation training in nursing students on their knowledge, skills, satisfaction and self-confidence levels, it was planned to be performed in a randomized controlled type.

The population of the research will be 4th grade students enrolled in the Faculty of Health Sciences, Faculty of Nursing . The sample of the study will consist of all 4th grade students who meet the sample selection criteria.

Sampling Inclusion Criteria: Individuals over the age of 18, who agreed to participate in the study in written and verbal form, and participated in all phases of the study will be included.

In the randomization part of the study, the students will assigned to the experiment (n=30) and control (n=30) groups according to their number in the class list using the random numbers table.

Data will collect with "Sociodemographic Data Form", "Cardiopulmonary Resuscitation Knowledge Test", "Cardiopulmonary Resuscitation Skills Checklist" and "Student Satisfaction and Confidence in Learning Scale".

Written permission will be obtained from the individuals who volunteered to participate in the study, and "Sociodemographic Data Form" and "Cardiopulmonary Resuscitation Knowledge Test" will be applied to all students.

Cardiopulmonary Resuscitation training will be given theoretically to all students in the classroom environment by an expert academician who has an associate professor in the field of Surgical Nursing. This training will take 1 hour.

The names of all students will be written in alphabetical order, and students will be divided into "Haptic" or "Highly Fidelity Simulator" groups using the random numbers table.

Intervention in Haptic Group: Students will perform Cardiopulmonary resuscitation using 3D Systems Touch Haptic Simulator. During the intervention, there will be 2 researchers and the student who made the application in the room. While one of the researchers will be with the student only for support during the practice, the other researcher will fill the "Cardiopulmonary Resuscitation Skills Checklist" by evaluating the cardiopulmonary resuscitation skill of the student.

Intervention in the High Fidelity Simulator Group: Students will perform Cardiopulmonary resuscitation using High Fidelity CPR Simulator. During the intervention, there will be 2 researchers and the student who made the application in the room. While one of the researchers will be with the student only for support during the practice, the other researcher will fill the "Cardiopulmonary Resuscitation Skills Checklist" by evaluating the cardiopulmonary resuscitation skill of the student. The application of the student will take a total of 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Over18 years old
* Being 4nd year student
* Volunteering to take a CPR training
* who agreed to participate in the study in written and verbal form,
* participated in all phases of the study will be included.

Exclusion Criteria:

* Not being volunteer to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-02 (Estimated); Primary Completion 2022-08-02 (Estimated); Study Completion 2022-10-02 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic Data of the students | Baseline
  The form in which the socio-demographic data of the students such as age and gender are questioned.
Change from Resuscitation Knowledge Test at 3 weeks | Baseline and 3 week later.
  Using the books, articles and guides in the literature, 15 multiple-choice questions about CPR were prepared and will be measured with the Resuscitation Knowledge Test. The maximum score to be obtained from this test is 15 and the minimum 0.
Cardiopulmonary Resuscitation Skills Checklist | after 1 hour of CPR training (while the student is practicing CPR skill)
  While practicing, the student will be evaluated by the observer with a 20-step checklist. Each step will be evaluated as "applied", "partially implemented", "not implemented". The highest score is 100, the lowest score is 0.

SECONDARY OUTCOMES:
Student Satisfaction and Self-Confidence in Learning Scale | within 10 minutes, after the student has practiced the CPR skill
  This instrument is a 12-item scale. It has 2 sub-dimensions: "Satisfaction with current learning"(5 items) and "Self-Confidence in Learning"(7 items).
  Responses are rated on a 5-point Likert scale with values ranging from 1 (strongly disagree) to 5 (strongly agree).
  The highest score is 60, the lowest score is 12. It is evaluated that as the score increases, student satisfaction and self-confidence in learning increase.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Kabuk, PhD, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
If it is necessary for the ethical issue, investigators can share.

REFERENCES:
- [Result] Panchal AR, Berg KM, Hirsch KG, Kudenchuk PJ, Del Rios M, Cabanas JG, Link MS, Kurz MC, Chan PS, Morley PT, Hazinski MF, Donnino MW. 2019 American Heart Association Focused Update on Advanced Cardiovascular Life Support: Use of Advanced Airways, Vasopressors, and Extracorporeal Cardiopulmonary Resuscitation During Cardiac Arrest: An Update to the American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2019 Dec 10;140(24):e881-e894. doi: 10.1161/CIR.0000000000000732. Epub 2019 Nov 14. PMID 31722552
- [Result] Su XH, Deng Z, He BW, Liu YQ. Haptic-based virtual reality simulator for lateral ventricle puncture operation. Int J Med Robot. 2020 Dec;16(6):1-10. doi: 10.1002/rcs.2176. Epub 2020 Oct 12. PMID 32991775
- [Result] Unver V, Basak T, Watts P, Gaioso V, Moss J, Tastan S, Iyigun E, Tosun N. The reliability and validity of three questionnaires: The Student Satisfaction and Self-Confidence in Learning Scale, Simulation Design Scale, and Educational Practices Questionnaire. Contemp Nurse. 2017 Feb;53(1):60-74. doi: 10.1080/10376178.2017.1282319. Epub 2017 Feb 10. PMID 28084900
- [Result] Winship C, Williams B, Boyle MJ. Cardiopulmonary resuscitation before defibrillation in the out-of-hospital setting: a literature review. Emerg Med J. 2012 Oct;29(10):826-9. doi: 10.1136/emermed-2011-200080. Epub 2011 Nov 22. PMID 22109533
- See also: TURKISH CARDIOLOGY ASSOCIATION — http://tkd.org.tr/ileri-kardiyak-yasam-destegi-kursu/sayfa/tyd